CLINICAL TRIAL: NCT06902415
Title: Research on the Application of Quantitative Digital Subtraction Angiography Hemodynamic Analysis Platform in Cerebrovascular Diseases
Brief Title: Application of QDSA Platform in Cerebrovascular Diseases
Acronym: RADAR
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024-371-02
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cerebrovascular Disease
Keywords: Cerebrovascular Disease; Quantitative Digital Subtraction Angiography; Hemodynamic; Stroke; Death; Outcome
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Testing populations: Patients with cerebrovascular disease can be evaluated for quantitative hemodynamic characteristics using QDSA.
  Interventions: Device: QDSA (Quantitative Digital Subtraction Angiography)

INTERVENTIONS:
Device: QDSA (Quantitative Digital Subtraction Angiography) — QDSA is a quantitative analysis technology based on DSA, used to assess hemodynamic characteristics and provide critical data support for the diagnosis and treatment of cerebrovascular diseases.

SUMMARY:
Cerebrovascular diseases pose a major global public health challenge, characterized by exceptionally high mortality and disability rates, with their pathogenesis closely linked to hemodynamic abnormalities. The quantitative digital subtraction angiography (QDSA) analysis platform, leveraging its advantages of vessel modeling-free operation, high computational efficiency, and DSA-equivalent sensitivity, has emerged as a novel hemodynamic assessment method with significant clinical potential. This study aims to establish a cerebrovascular disease cohort incorporating QDSA parameters to systematically validate the clinical value of this technology in preoperative evaluation and surgical planning, thereby providing evidence-based insights for optimizing diagnostic and therapeutic strategies.

DETAILED DESCRIPTION:
Study overview: This study will construct a prospective cohort dataset that comprehensively integrates DSA features, clinical baseline data, clinical manifestations, and follow-up data. Using QDSA technology, hemodynamic parameters of patients will be extracted. Based on multidimensional data, this study will conduct clinical research targeting different clinical scenarios, covering disease natural history evaluation, risk factor analysis, and treatment efficacy assessment. Through longitudinal tracking of data evolution and multidimensional parameter correlation analysis, this framework aims to establish an evidence-based pathway for translating hemodynamic characteristics into clinical decision-making, providing valuable references for clinical practice.

Sample size: Between February 2025 and February 2030, a total of 1000 patients with cerebrovascular diseases will be prospectively enrolled, including those with cerebral arteriovenous malformations (AVMs), cerebral aneurysms, moyamoya disease, cerebral arterial stenosis, ischemic stroke, and other subtypes.

Study endpoints: The primary outcome is defined as the composite endpoint of symptomatic stroke or death. And the secondary outcome included neurological status, assessed using the modified Rankin Scale (mRS).

Follow-up: Follow-up assessments will be conducted at 3 months, 6 months, annually (1 year, 2 years, and 3 years), and every 5 years after the initial treatment decision in the form of telephone interviews or record review. Individuals suspected of experiencing cerebrovascular events will undergo focused documentation during each telephone contact or record review.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebrovascular diseases diagnosed and assessed by DSA for related risks and treatment options.
2. The DSA acquisition protocol complies with the standard procedure.
3. DSA images must include complete anteroposterior and lateral views.
4. Raw data must be available in DICOM format.
5. Image quality and pixel resolution must support data analysis.
6. Patients must undergo regular follow-ups.

Exclusion Criteria:

1. Cerebrovascular diseases not diagnosed or risk-assessed using DSA.
2. Patients with DSA image quality insufficient for image analysis and processing.
3. Severe organ diseases with an expected survival period of less than 2 years.
4. Inability to cooperate with treatment and follow-up.
5. Participation in other clinical trials within the past 6 months.
6. Other conditions deemed by the investigator as unsuitable for participation in this trial.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebrovascular disease can be evaluated for quantitative hemodynamic characteristics using QDSA.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Symptomatic stroke or death | After treatment (max 10 years)
  Stroke is defined as a clinically symptomatic event (any new focal neurological deficit, seizure, or new-onset headache) that is associated with imaging findings of hemorrhage or infarction. Hemorrhage is defined as fresh intracranial blood on head computed tomography (CT) or magnetic resonance imaging (MRI), or in the cerebrospinal fluid. Infarction is defined as a new ischemic lesion on cranial CT or MRI (diffusion-weighted, T2-weighted, or fluid-attenuated inversion recovery MRI).

SECONDARY OUTCOMES:
Neurological status (modified Ranking Scale score) | After treatment (max 10 years)
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided